CLINICAL TRIAL: NCT01008670
Title: Identification of the Pericardiophrenic Vein During Cardiac Device Implant Procedures to Prevent Extracardiac Stimulation
Acronym: IDPV-003
Status: Completed | Type: Observational
Sponsor: Respicardia, Inc. (Industry)
Responsible Party: Lori Austin, Cardiac Concepts, Inc.
Other Study IDs: CCI-Venography
Record Dates: First submitted 2009-11-04; First posted 2009-11-06 (Estimated); Last update posted 2010-11-24 (Estimated); Status verified 2010-11

CONDITIONS: Heart Failure
Keywords: Cardiac resynchronization therapy
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Device Implant Recipients: Patients undergoing CRT implantation, or candidates for future CRT devices currently undergoing ICD or pacemaker implantation.

SUMMARY:
The primary goal of this study is to develop techniques to identify the course of the phrenic nerve in patients already undergoing cardiac resynchronization therapy (CRT) implantation or candidates for future CRT devices undergoing implantable cardioverter-defibrillator (ICD) or pacemaker implantation. Specifically, the study intends to identify the location and course of the left pericardiophrenic vein, and thus the left phrenic nerve, to guide the location for coronary vein lead placement and minimize the risk of phrenic nerve stimulation.

DETAILED DESCRIPTION:
Phrenic nerve stimulation from cardiac resynchronization therapy (CRT) is a common adverse event occurring in 1.5-3% of patients and sometimes as high as 10%. Phrenic nerve stimulation is frequently observed during the implantation procedure but often appears shortly after implantation as well. Clinically, dyspnea, cough, and hiccups can occur, some of which are uncomfortable and not tolerated by the patient for very long periods of time. Resolution of these clinical outcomes requires repositioning the left coronary vein lead in a second procedure with its attendant serious clinical sequelae. As CRT leads become smaller the incidence of phrenic nerve stimulation is likely to increase.

The risk of phrenic nerve stimulation (PNS) exists during CRT implantation and is only minimally dependent of the type of coronary lead and highly dependent upon location of the left coronary vein lead in relationship to the left phrenic nerve and stimulation strength. Tedrow et al. demonstrated in a cohort of 71 patients PNS can reach 16% if stimulation strength is increased to maximize mechanical benefit of CRT. No current methods have been able to predict PNS, the one likely method of preventing PNS is to identify the location of the phrenic nerve in the specific patient, as confirmed by visualization and ability to stimulate the phrenic nerve and by maximizing the distance between the coronary vein lead position and nerve.

In order to reduce the incidence of phrenic nerve stimulation, Vaseghi performed non-selective injections of contrast media and was able to identify the left pericardiophrenic vein in only about 12% of patients undergoing biventricular pacemaker placement. However, in these patients, identification of the left pericardiophrenic vein provides a landmark for positioning of the left ventricular (LV) lead that totally eliminated the incidence of phrenic nerve pacing.

The relationship of cardiac structures to the right and left phrenic nerves is generally known but is significantly variable between patients. There is no imaging or other clinically available modality that allows the physician to identify the location of the left phrenic nerve and attempt to avoid it during the left coronary vein lead implant procedure.

The pericardiophrenic veins are a deep collateral venous drainage of the pericardium, pleura and diaphragm and lie adjacent the phrenic nerves on both the right and left sides between the parietal pericardium and adjacent pleura. The ostium of the left pericardiophrenic vein is usually in the left brachiocephalic vein opposite the entrance of the left jugular vein. The left phrenic vein is located in the general vicinity of the thymic veins which often have multiple ostia in close proximity. There are several case reports in the literature of inadvertent cannulation of the pericardiophrenic veins with Swan-Ganz catheters, central venous catheters and one report of cannulation with a pacing lead leading to inadvertent phrenic nerve pacing.

The primary goal of this study is to develop techniques to identify the course of the phrenic nerve in patients already undergoing cardiac resynchronization therapy (CRT) implantation or candidates for future CRT devices undergoing implantable cardioverter-defibrillator (ICD) or pacemaker implantation. Specifically, the study intends to identify the location and course of the left pericardiophrenic vein, and thus the left phrenic nerve, to guide the location for coronary vein lead placement and minimize the risk of phrenic nerve stimulation.

ELIGIBILITY:
Inclusion Criteria:

* Male or female between the ages of 18 and 85 years old.
* Undergoing implantation of a CRT, ICD, or pacemaker device

Exclusion Criteria:

* Allergy to contrast dye
* Nursing mothers and women who are pregnant
* Patients for whom informed consent cannot be obtained.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients currently under the care of an electrophysiologist or cardiac device implanter who are scheduled to receive a CRT device, or those patients receiving an ICD or pacemaker device who are future candidates for CRT device implantation.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2007-12; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
The primary endpoint of this study is to determine if methods can be developed for identifying the course of the left vein, thus the location of the phrenic nerve, during a device implant procedure. | Methods are assessed acutely (during the lead implant procedure)

CONTACTS AND LOCATIONS:
Locations (13):
- United States (6):
  - University of Alabama, Birmingham, Alabama
  - Johns Hopkins University, Baltimore, Maryland
  - Ohio Heart Hospital, Cincinnati, Ohio
  - The Ohio State University, Columbus, Ohio
  - Baptist Memorial Hospital, Nashville, Tennessee
  - Sentara Norfolk General, Norfolk, Virginia
- Germany (2):
  - Ruhr University of Bochum, Bad Oeynhausen
  - University of Mannheim, Mannheim
- Prince of Wales Hospital, Shatin, New Territories, Hong Kong
- Policlinico di Monza, Monza, Italy
- Poland (3):
  - Jagiellonian University, Krakow
  - Medical Military Institute, Warsaw
  - Wroclaw Fourth Military Hospital, Wroclaw